CLINICAL TRIAL: NCT01236066
Title: A Study on the Impact of Rotavirus Vaccination on Hospitalisations for Rotavirus Gastroenteritis in Children Aged <5 Years in Australia
Brief Title: Impact of Rotavirus Vaccination on Hospitalisations for Rotavirus Gastroenteritis in Children Aged <5 Years in Australia
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 114910
Record Dates: First submitted 2010-10-28; First posted 2010-11-08 (Estimated); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Rotavirus Gastroenteritis; Gastroenteritis
Keywords: Rotavirus Gastroenteritis; Rotarix; RotaTeq; Gastroenteritis
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Study Group: Australian children aged < 5 years who have been vaccinated with RotaTeq or Rotarix from 2007 to 2009 as well as all children aged < 5 years hospitalised for all-cause gastroenteritis, rotavirus gastroenteritis or bronchiolitis.
  Interventions: Other: Database analysis

INTERVENTIONS:
Other: Database analysis — Existing computerised administrative databases from the Australian Institute of Health and Welfare (AIHW) will be reviewed to retrieve data on all-cause gastroenteritis/ rotavirus enteritis and bronchiolitis hospitalisations of children <5 years in all the states using Rotarix from 1998 to 2009. Data from Australian Childhood Immunisation Register (ACIR) post introduction of rotavirus vaccines in the National Immunisation Program (2007 to 2009) will also be used.

SUMMARY:
This study aims to monitor the incidence rates and duration of hospitalisations for rotavirus gastroenteritis (RV GE) and all cause GE, compared to bronchiolitis from 1998 to 2009, in children < 5 years of age after the introduction of Rotarix in 2006 by year, both inside and outside rotavirus season in Australia. It further aims to compare the two dose regimen of Rotarix with the three dose regimen of RotaTeq from 2007 to 2009.

ELIGIBILITY:
Inclusion Criteria:

* Children <5 years of age;
* Children with a diagnosis of all-cause gastroenteritis, rotavirus gastroenteritis or bronchiolitis in the Australian Institute of Health and Welfare (AIHW) database in New South Wales, Australian Capital Territory, Tasmania and Northern Territory, from 1998 to 2009;
* Children who were vaccinated with Rotarix or RotaTeq in New South Wales and Queensland, registered in the Australian Childhood Immunisation Register (ACIR) database in Queensland and New South Wales, from 2007 to 2009.

Exclusion Criteria:

No exclusion criteria will be applied.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Australian children aged < 5 years who have been vaccinated with RotaTeq (in Queensland) and Rotarix (in New South Wales) from 2007 to 2009 as well as all children aged < 5 years hospitalised for all-cause gastroenteritis, rotavirus gastroenteritis or bronchiolitis, before and after introduction of Rotarix vaccination in New South Wales, Australian Capital Territory, Tasmania and Northern Territory, from 1998 to 2009.
Sampling Method: Non-Probability Sample
Enrollment: 1 (Actual)
Dates: Start 2010-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Occurrence of all cause gastroenteritis (GE) in children < 5 years by age group, state and year | Each year: 1998, 1999, 2000, 2001, 2002, 2003, 2004, 2005, 2006, 2007, 2008, 2009
Occurrence of rotavirus gastroenteritis (RV GE) in children < 5 years by age group, state and year | Each year: 1998, 1999, 2000, 2001, 2002, 2003, 2004, 2005, 2006, 2007, 2008, 2009
Occurrence of bronchiolitis in children < 5 years by age group, state and year | Each year: 1998, 1999, 2000, 2001, 2002, 2003, 2004, 2005, 2006, 2007, 2008, 2009
Mean age of full immunisation of Rotarix and RotaTeq in New South Wales and Queensland | From 2007 to 2009
Percentage of full immunisation of Rotarix and RotaTeq in New South Wales and Queensland according to age-specific recommendations for rotavirus (RV) immunisation in Australia | From 2007 to 2009
Percentage of full immunisation of Rotarix and RotaTeq in New South Wales and Queensland outside of age-specific recommendations for rotavirus (RV) immunisation in Australia | From 2007 to 2009
Percentage of children immunised with the last dose of Rotarix according to age-specific recommendations for rotavirus (RV) immunisation in Australia | From 2007 to 2009
Percentage of children immunised with the last dose of Rotarix outside of age-specific recommendations for rotavirus (RV) immunisation in Australia | From 2007 to 2009
Percentage of children immunised with the last dose of RotaTeq according to age-specific recommendations for rotavirus (RV) immunisation in Australia | From 2007 to 2009
Percentage of children immunised with the last dose of RotaTeq outside of age-specific recommendations for rotavirus (RV) immunisation in Australia | From 2007 to 2009

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline

REFERENCES:
- [Derived] Pendleton A, Galic M, Clarke C, Ng SP, Ledesma E, Ramakrishnan G, Liu Y. Impact of rotavirus vaccination in Australian children below 5 years of age: a database study. Hum Vaccin Immunother. 2013 Aug;9(8):1617-25. doi: 10.4161/hv.24831. Epub 2013 Jun 3. PMID 23733041